CLINICAL TRIAL: NCT00182728
Title: Partial Breast Treatment Using Single Dose Intraoperative Radiotherapy for Patients With Early Stage Breast Cancer - A Feasibility Study With Molecular Analysis of Tumors and Normal Breast Epithelial Tissue
Brief Title: Radiation Therapy During Surgery in Treating Older Women With Invasive Breast Cancer
Acronym: NRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0218
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast | interventions — Surgical Procedures, Operative; Therapeutics; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative Radiation Arm (Experimental): Intraoperative radiotherapy (radiation therapy) during surgery for tumor excision.
  Interventions: Procedure: surgery; Procedure: therapy; Radiation: radiation therapy

INTERVENTIONS:
Procedure: surgery — conventional
Procedure: therapy — neoadjuvant
Radiation: radiation therapy — intraoperative radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation during surgery may be an effective treatment for breast cancer.

PURPOSE: This phase II trial is studying how well radiation therapy works in treating older women who are undergoing surgery for invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of intraoperative partial breast radiotherapy prior to surgical resection in older women with low-risk early stage primary invasive ductal carcinoma of the breast. Feasibility will be determined by the rate of good/excellent cosmesis, as measured by the Radiation Therapy Oncology Group (RTOG) cosmetic rating scale, in patients treated with this regimen compared with that of patients treated with partial breast brachytherapy in clinical trial RTOG-9517.
* Determine the incidence of grade 3-4 toxicity of this regimen in these patients.
* Determine the rate of ipsilateral breast recurrence, including recurrence within the tumor bed as compared to elsewhere in the breast, in patients treated with this regimen.

Secondary

* Determine the radiation-induced activation of receptors and signal transduction pathways involved in radiation response in patients treated with this regimen.

OUTLINE: This is a non-randomized study.

Patients undergo intraoperative lymphatic mapping and sentinel lymphadenectomy OR standard level I, II axillary dissection to evaluate the lymph nodes followed by intraoperative breast ultrasonography to define the tumor target volume. Patients then undergo intraoperative single-dose partial breast radiotherapy followed by segmental mastectomy (i.e., lumpectomy) of the tumor. Patients with 1 or 2 tumor-involved surgical margins may undergo repeat segmental mastectomy. Patients with > 2 tumor-involved surgical margins undergo mastectomy. Patients determined to have a tumor size > 3 cm or an extensive intraductal component on final pathology evaluation undergo standard external beam radiotherapy after surgery.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 71 patients will be accrued for this study within 2 to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive ductal carcinoma of the breast

  * Tumor size ≤ 3 cm
  * No extensive intraductal component
  * Tumor must not be attached to the skin, underlying muscle, or chest wall
* Candidate for breast-conserving therapy, as determined by the surgical and radiation oncologist

  * Tumor amenable to segmental mastectomy (i.e., lumpectomy)
* No bilateral breast cancer
* No clinical or radiographic multifocal disease not amenable to single segmental mastectomy

  * Patients with > 1 tumor mass in the same breast must have only 1 mass that is histologically malignant AND all other masses must be proven histologically benign
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 48 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* 0-2

Life expectancy

* At least 5 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* Fertile patients must use effective contraception
* No collagen vascular disease
* No medical condition that would preclude surgery
* Other prior malignancy allowed provided the following criteria are met:

  * Patient has undergone potential curative therapy for all prior malignancies
  * There is no evidence of any prior malignancy within the past 5 years
  * Patient is deemed to be at low risk for recurrence of prior malignancy, as determined by the treating physician

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for this malignancy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the breast

Surgery

* No breast implants

Ages: 48 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-03-18 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2019-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Olilla, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Ollila DW, Klauber-DeMore N, Tesche LJ, Kuzmiak CM, Pavic D, Goyal LK, Lian J, Chang S, Livasy CA, Sherron RF, Sartor CI. Feasibility of breast preserving therapy with single fraction in situ radiotherapy delivered intraoperatively. Ann Surg Oncol. 2007 Feb;14(2):660-9. doi: 10.1245/s10434-006-9154-1. PMID 17091330
- [Background] Stitzenberg KB, Klauber-Demore N, Chang XS, Calvo BF, Ollila DW, Goyal LK, Meyers MO, Kim HJ, Tepper JE, Sartor CI. In vivo intraoperative radiotherapy: a novel approach to radiotherapy for early stage breast cancer. Ann Surg Oncol. 2007 Apr;14(4):1515-6. doi: 10.1245/s10434-006-9152-3. PMID 17235715
- [Result] Kimple RJ, Klauber-DeMore N, Kuzmiak CM, Pavic D, Lian J, Livasy CA, Chiu WM, Moore DT, Sartor CI, Ollila DW. Local control following single-dose intraoperative radiotherapy prior to surgical excision of early-stage breast cancer. Ann Surg Oncol. 2011 Apr;18(4):939-45. doi: 10.1245/s10434-010-1392-6. PMID 21061074
- [Result] Vanderwalde NA, Jones EL, Kimple RJ, Moore DT, Klauber-Demore N, Sartor CI, Ollila DW. Phase 2 study of pre-excision single-dose intraoperative radiation therapy for early-stage breast cancers: six-year update with application of the ASTRO accelerated partial breast irradiation consensus statement criteria. Cancer. 2013 May 1;119(9):1736-43. doi: 10.1002/cncr.27915. Epub 2013 Jan 29. PMID 23361892
- [Result] Kimple RJ, Klauber-DeMore N, Kuzmiak CM, Pavic D, Lian J, Livasy CA, Esler L, Moore DT, Sartor CI, Ollila DW. Cosmetic outcomes for accelerated partial breast irradiation before surgical excision of early-stage breast cancer using single-dose intraoperative radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):400-7. doi: 10.1016/j.ijrobp.2009.10.032. Epub 2010 Apr 13. PMID 20395062
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2003 to July 2007
Pre-assignment Details: 89 patients consented. Of those 89, 18 were not treated for the following reasons: tumor not seen on ultrasound (2), tumor too close to chest wall (7), tumor too large (1), ineligible pathology (1), ineligible nodal status (1), operating room logistical errors (3), patients withdrew (2), not eligible for anesthesia (1).
Period: Overall Study
Arm/Group | Intraoperative Radiation Arm
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 71
Age, Continuous [Mean (Full Range); unit: years] | 64.8 [48 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71
Clinical Staging [Count of Participants; unit: Participants] — The TNM Classification of Malignant Tumours (TNM) is a cancer staging notation system that describes the stage of a cancer which originates from a solid tumor with alphanumeric codes. Higher numbers mean the cancer is more advanced.
  T describes the size of the original (primary) tumor and whether it has invaded nearby tissue, N describes nearby (regional) lymph nodes that are involved, M describes distant metastasis (spread of cancer from one part of the body to another).
  Participants
    cT1a | 2
    cT1b | 18
    cT1c | 35
    cT2 (<3 cm) | 16
    cN0 | 71
Grade [Count of Participants; unit: Participants] — Tumor grade is the description of a tumor based on how abnormal the tumor cells and the tumor tissue look under a microscope. It is an indicator of how quickly a tumor is likely to grow and spread. The grading system is as follows: grade I - cancer cells that resemble normal cells and aren't growing rapidly. grade II - cancer cells that don't look like normal cells and are growing faster than normal cells. grade III - cancer cells that look abnormal and may grow or spread more aggressively
  Participants
    I | 25
    II | 24
    III | 22
Markers [Count of Participants; unit: Participants] — Tumor markers are substances that are produced by cancer or by other cells of the body in response to cancer or certain benign (noncancerous) conditions. The following markers are proteins.
  Participants
    Estrogen Receptor (ER) positive | 54
    Progesterone Receptor (PR) positive | 50
    Human Epidermal Growth Factor receptor (HER) 2 pos | 8
    ER+, PR+, HER2- | 46
    "triple negative" | 12

OUTCOME MEASURES:

1. Primary Outcome: Rates of Good/Excellent Cosmesis as Measured by the Radiation Therapy Oncology Group (RTOG) Cosmetic Rating Scale - Rated by Physician
Description: Rates of good/excellent cosmesis was evaluated using the following criteria:
  Excellent - when compared to the untreated breast, there is minimal or no difference in the size, shape, or texture of the treated breast. There may be mild thickening or scar tissue within the breast or skin, but not enough to change the appearance.
  Good - there is mild asymmetry in the size or shape of the treated breast as compared to the normal breast. The thickening or scar tissue within the breast causes only a mild change in the shape.
Time Frame: 1 year follow up visit
Population: Patients who received intraoperative radiation therapy (IORT) alone. 56 patients were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 56
Participants | 45

2. Primary Outcome: Rates of Good/Excellent Cosmesis as Measured by the Radiation Therapy Oncology Group (RTOG) Cosmetic Rating Scale - Rated by Patients
Description: as for outcome 1
Time Frame: 1 year follow up visit
Population: Patients who received IORT alone. 42 patients assessed their cosmetic outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 42
Participants | 32

3. Primary Outcome: Incidence of Grade 3/4 Toxicity
Description: Skin and subcutaneous toxicity were graded by a radiation oncologist according to the common terminology criteria for adverse events version 3.0. Toxicities directly, probably, or possibly related to the radiation were included. Grade refers to the severity of the AE. The CTCAE v3.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each adverse event (AE) based on this general guideline:
  Grade 1 Mild Adverse Event Grade 2 Moderate Adverse Event Grade 3 Severe Adverse Event Grade 4 Life-threatening or disabling Adverse Event Grade 5 Death related to Adverse Event
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 71
Participants | 0

4. Primary Outcome: Ipsilateral Breast Recurrence
Description: Percentage of participants who experienced a ipsilateral breast event (tumor bed recurrence versus elsewhere in breast).
Time Frame: 5 years
Population: There were 71 patients who received IORT. Of those 71 patients, 18 received further local therapy due to "high risk" pathology. The results include the 53 patients who received IORT without further local therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 53
percentage of participants | 13 [6 to 26]

5. Secondary Outcome: Association of Phosphorylated Epidermal Growth Factor Receptor (EGFR) , Human Epidermal Growth Factor Receptor 2 (HER2), p44/42 Mitogen-activated Protein Kinase (MAPK), and Protein Kinase B (Akt) in Breast Tumors and Normal Tissue Before and After IORT
Time Frame: 3 months
Population: No data were collected for any of these biomarkers. Although samples were obtained from patients, they were never processed and analyzed.
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Association of Nuclear Factor Kappa-light-chain-enhancer of Activated B Cells (NFkB) Expression in Tumor and Normal Tissue Before and After IORT
Time Frame: 3 months
Population: No data were collected for this biomarker. Although samples were obtained from patients, they were never processed and analyzed.
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Association of Nuclear p53 Expression in Tumor and Normal Tissue Before and After IORT
Time Frame: 3 months
Population: as for outcome 6
Arm/Group | Intraoperative Radiation Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Acute toxicity was evaluated 1 week and 3 months after IORT
Arm/Group | Intraoperative Radiation Arm
All-Cause Mortality (participants affected / at risk) | 6/71
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 11/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Radiation Arm (N=71)
Alopecia (Skin and subcutaneous tissue disorders) | 1
Low blood counts (Blood and lymphatic system disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Congestive heart failure (CHF) (Cardiac disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Seroma (Injury, poisoning and procedural complications) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Edema: limb (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Intraoperative breast injury (Injury, poisoning and procedural complications) | 1
Myocardial infarction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Changes in vision (Eye disorders) | 1
Pain - Head/headache (Nervous system disorders) | 1
Skin (cellulitis) (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes